CLINICAL TRIAL: NCT01589224
Title: Risk Factor Analysis for Coronary Atherosclerosis Measured by MDCT
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: KoreaHealth_MDCT
Record Dates: First submitted 2012-04-24; First posted 2012-05-01 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-04

CONDITIONS: Atherosclerosis; Metabolic Syndrome
MeSH Terms: conditions — Atherosclerosis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy people

SUMMARY:
Coronary MDCT (multi-detector computed tomography) has been useful screening imaging modality for the coronary artery disease. Recently, novel adipokines and hepatokines as well as various inflammatory markers have been known as direct regulators of atherosclerosis. Therefore, the investigators examine the correlation of various metabolic risk factors including adipokines and hepatokines with coronary atherosclerosis measured by coronary MDCT in apparently healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy people who underwent medical routine check up in Korea Health Promotion Center.
* age > 20 years

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* Diabetes
* Stage 2 hypertension
* Severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy people who underwent medical routine check up in Korea Helath Promotion Center.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
relation of adipokines and hepatokines with coronary atherosclerosis measured by MDCT | 3month
  to examine the correlation of serum concentration of various adipokine such as adiponectin, resistin, A-FABP with coronary atheroslcerosis measured by MDCT as AGATSTON score, modified Gensini score

SECONDARY OUTCOMES:
relation of adipokines and hepatokines with coronary atherosclerosis measured by MDCT | 3months
  to examine the correlation of serum concentration of various hepatokines such as FGF-21, fetuin- A and selenoprotein P with coronary atheroslcerosis measured by MDCT as AGATSTON score, modified Gensini score
the correlation of various inflammatory markers with coronary atherosclerosis | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- korea University Guro Hospital, Seoul, South Korea